CLINICAL TRIAL: NCT06350721
Title: Feasibility, Usability and Safety of the Vestibular Rehabilitation Using the Immersive Virtual Reality Software DizzyVR
Acronym: DizzyVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Loyola Andalucia (Other)
Collaborators: University of Seville (Other); Universitat Politècnica de València (Other); Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Cristina García-Muñoz, Principal investigator, Universidad Loyola Andalucia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DizzyVR
Record Dates: First submitted 2024-01-17; First posted 2024-04-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Vestibular Disorder; Physical Disability
Keywords: Virtual reality; Vestibular; Head Mounted Display; DizzyVR
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Each patient will receive a total of 8 sessions of vestibular rehabilitation with the DizzyVR system. Each session will last for 50 minutes, with a frequency of one session per week. The total duration of the intervention will be 10 weeks, with the initial assessment/T0 taking place in the first week and the final assessment/T2 in the tenth week. Similarly, the total expected participation time for each participant is set at 12 weeks (T3).
  Interventions: Device: DizzyVR

INTERVENTIONS:
Device: DizzyVR — Each patient will receive a total of 8 sessions of vestibular rehabilitation with the DizzyVR system. Each session will last for 50 minutes, with a frequency of one session per week. The total duration of the intervention will be 10 weeks, with the initial assessment/T0 taking place in the first week and the final assessment/T2 in the tenth week. Similarly, the total expected participation time for each participant is set at 12 weeks (T3).

SUMMARY:
The main goals of this pilot study is to assess the feasibility, usability, satisfaction and safety of the immersive virtual reality system called DizzyVR in participants diagnosed with a vestibular disorder. In addition, it aims to collect preliminary data about clinical effectiveness. The main questions it aims to answer are:

* To assess the feasibility, usability and safety of the system DizzyVR for the vestibular rehabilitation in participants with vestibular disorders.
* To detect and record possible adverse events due to the use of DizzyVR.
* To examine the degree of adherence of the participants to the intervention.
* To know the average success rate of the different games in each session.
* To evaluate the average difficulty levels overcome throughout the intervention.
* To know the usability and satisfaction with the system reported by participants and therapists.
* To assess preliminary efficacy data on the impact of this new vestibular rehabilitation system on dizziness, gait speed, balance confidence and gait stability.

Participants will receive the vestibular rehabilitation based on the novel immersive virtual systema, DizzyVR.

DETAILED DESCRIPTION:
Once the patient is received in the physiotherapy area of the Vertigo Unit, the researchers will proceed to provide the informational sheet and informed consent, as well as verbally explain the project. After the informed consent is signed, the researchers will collect all descriptive variables, as well as the baseline score of the DHI questionnaire (T0). During the course of the research, the researchers will daily record participants' attendance, the overall percentage of correct answers in each session, the occurrence of undesired effects, and the score of the Simulator Sickness Questionnaire (T1). In the final physiotherapy session (T2), each participant will re-evaluate the DHI questionnaire, as well as the perceived usability questionnaire of the system (SUS) and the virtual systems satisfaction evaluation questionnaire (USEQ). Finally, approximately 15 days after the intervention concludes, participants will be scheduled for in-depth individual perceptions about the system through a semi-structured interview (T3). With the same purpose, after the period of using the DizzyVR system, the researchers will interview the physiotherapists who have participated in this study (T4).

Each patient will receive a total of 8 sessions of vestibular rehabilitation with the DizzyVR system. Each session will last for 50 minutes, with a frequency of one session per week. The total duration of the intervention will be 10 weeks, with the initial assessment/T0 taking place in the first week and the final assessment/T2 in the tenth week. Similarly, the total expected participation time for each participant is set at 12 weeks (T3).

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 75.
* Confirmed diagnosis of central or peripheral vestibulopathy.
* Preserved walking ability.
* Presence of dizziness symptoms as assessed by the Dizziness Handicap Inventory (> 10 points).

Exclusion Criteria:

* Severe visual impairments.
* Cognitive impairment (Mini Mental State Examination < 24).
* Existence of comorbidities severely affecting postural control and balance.
* Uncontrolled systemic diseases that contradict physical activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence rate | 10 weeks
  percentage of completed sessions
Success rate | 10 weeks
  Mean success rates of the games per session
Progression | 10 weeks
  Levels of the games accomplished during the sessions.
System Usability Scale (SUS) | 10 weeks
  Participants perceived usability of the system.
User Satisfaction Evaluation Questionnaire (USEQ) | 10 weeks
  Acceptability of the prototype device/software
Simulator Sickness Questionnaire (SSQ) | 10 weeks
  Security of the system
Register of risk and number of adverse events experimented by the stakeholders | 10 weeks
  Security of the prototype device

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | 10 weeks
  Dizziness symptoms
Timed Up and Go Test (TUG) | 10 weeks
  Gait speed
Activities-specific Balance Confidence Scale (ABC) | 10 weeks
  Perceived balance confidence
Functional Gait Assessment questionnaire (FGA) | 10 weeks
  Gait stability

CONTACTS AND LOCATIONS:
Overall Officials: MARIA JESÚS CASUSO-HOLGADO, PhD, Principal Investigator — University of Seville
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Data of study will be only manage by the researchers of study and the physiotherapist of the clinic